CLINICAL TRIAL: NCT05798923
Title: A Phase 2a Single-Arm, Open-Label, Exploratory Study to Assess the Effects of LAM-001 for the Treatment of Pulmonary Hypertension
Brief Title: A Phase 2a Study of LAM-001 for the Treatment of Pulmonary Hypertension
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM-001-PAH-CLN01
Record Dates: First submitted 2023-03-13; First posted 2023-04-05 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LAM-001 (Experimental)
  Interventions: Drug: LAM-001

INTERVENTIONS:
Drug: LAM-001 — LAM-001 administered via dry powder inhalation

SUMMARY:
This is a clinical trial to assess the efficacy and safety of LAM-001 as an add-on therapy for the treatment pulmonary hypertension.

DETAILED DESCRIPTION:
This is a Phase 2a, single-arm, open-label, exploratory study assessing the efficacy and safety of LAM-001 as an add-on therapy for the treatment of WHO functional class III subjects with WSPH Group-1 or Group-3 pulmonary hypertension.

Approximately fifteen participants will receive standard of care plus LAM-001 once daily for the first 24 weeks of the study (Core Study).

Participants who complete the first 24 weeks on treatment and appear to have a favorable benefit-risk profile will be eligible to continue receiving LAM-001 for the remainder of the study (Extension Period) up to 12 months.

All participants will complete evaluations during a Follow-Up Period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Screening consistent with a diagnosis of precapillary PH (mPAP > 25 mmHg, PCWP < 18 mmHg, PVR >4WU) that is due to either:

   1. WSPH Group 1 PH (i.e., PAH of any of the following subtypes)

      * Idiopathic PAH
      * Heritable PAH
      * Drug- or toxin-induced PAH
      * PAH associated with connective tissue disease
      * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following shunt repair
   2. Confirmed diagnosis of WSPH Group 3 PH with advanced lung disease as defined by CT imaging (see Section 5.3.1) within 6- months of screening that demonstrates diffuse parenchymal lung disease or FVC < 65% of predicted for this cohort only, associated with one of the following:

   i. Idiopathic interstitial pneumonia (IIP) including:
   * Idiopathic pulmonary fibrosis (IPF)
   * Idiopathic nonspecific interstitial pneumonia
   * Respiratory bronchiolitis-associated interstitial ling disease (RB-ILD)
   * Unclassifiable idiopathic interstitial pneumonia ii. Chronic hypersensitivity pneumonitis (CHP) iii. Occupational lung disease (drug or radiation-induced) iv. Combined pulmonary fibrosis and emphysema (CPFE)
3. Symptomatic pulmonary hypertension classified as WHO functional class III
4. Pulmonary function tests within 6 months prior to Screening as follows:

   * For patients with WSPH Group 3 PH, forced vital capacity (FVC <65% predicted and a DLCO >30) for patients with confirmatory high- resolution computed tomography (CT) indicating fibrotic lung disease; For patients with WSPH Group 1 PAH, FVC ≥ 65%
   * For subjects with a history of lobectomy or pneumonectomy, and for whom there are no population-based normalization methods, assessment based on residual lung volume will be permitted to assess eligibility.
5. Ventilation-perfusion (VQ) scan, a CT pulmonary angiogram (CTPA) or pulmonary angiography, with findings that rule out chronic thromboembolic pulmonary hypertension. Can be performed any time prior to Screening or conducted during the Screening Period.
6. 6MWD ≥ 100 and ≤ 550 meters repeated twice during Screening Period and both values within 15% of each other, calculated from the highest value.
7. On a standard of care PAH therapy at stable (per SOC) dose levels for at least 30 days prior to screening. No SOC is required for Group 3 subjects but if on any therapy, this too should be stable for 30 days

   * For definition of SOC, see Section 5.1.1 Standard of Care
   * Stable dose is defined as no change in dose
8. Females of childbearing potential must satisfy following (details outlined in appendix, under Contraceptive Guidance and Collection of

   Pregnancy Information):
   1. Have 2 negative pregnancy tests as verified by the investigator prior to starting study and must agree to ongoing pregnancy testing during the study and at end of study treatment.
   2. If sexually active, must have used, and agree to continue to use, highly effective contraception without interruption, for at least 30 days prior to starting investigational product (IP), during the study (including dose interruptions), and for 90 days after discontinuation of study treatment.
   3. Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 90 days after the last dose of study treatment.
9. Male participants must:

   1. Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made from natural (animal) membrane (for example, polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 90 days following IP discontinuation, even if he has undergone a successful vasectomy.
   2. Refrain from donating sperm for the duration of the study and for 90 days after the last dose of study treatment.
10. Ability to adhere to the study visit schedule and understand and comply with all protocol requirements.
11. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Started or stopped receiving any general supportive therapy for pulmonary hypertension within 30 days prior to Week 0 Visit
2. Received IV inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to Week 0 Visit
3. History of atrial septostomy within 180 days prior to Screening Visit
4. History of more than moderate obstructive sleep apnea that is untreated
5. Prior exposure to oral sirolimus or any other mTOR inhibitor within last three months
6. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to Week 0 Visit or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible)
7. Uncontrolled systemic hypertension as evidenced by sitting systolic BP > 160 mmHg or sitting diastolic BP > 100 mmHg during Screening Visit after a period of rest
8. Systolic BP < 90 mmHg during Screening Visit or at baseline
9. History of known pericardial constriction
10. RHC contraindicated during the study per investigator
11. Personal or family history of long QTc syndrome or sudden cardiac death
12. Cerebrovascular accident within 3 months of Week 0 Visit
13. History of restrictive or constrictive cardiomyopathy
14. Left ventricular ejection fraction < 45% on echocardiogram performed within 6 months prior to Screening Period (or done as a part of the Screening Period), or PCWP > 18 mmHg as determined in the Screening Period RHC
15. Any current symptomatic coronary disease (myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain in the past 6 months prior to Screening Visit)
16. Acutely decompensated left or right heart failure within 30 days prior to Week 0 Visit, as per investigator assessment
17. Known diagnosis (as determined by echocardiography) of significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
18. Any of the following clinical laboratory values during the Screening Period prior to Week 0 Visit:

    1. Baseline Hgb > 16.0 g/dL within 28 days of Week 0 Visit
    2. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 3x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN within 28 days of Week 0 Visit
    3. Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (4-variable Modification of Diet in Renal Disease equation) within 28 days of Week 0 Visit or required renal replacement therapy within 90 days
19. History of opportunistic infection (e.g., invasive candidiasis or Pneumocystis pneumonia) within 6 months prior to Screening; serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to Screening
20. History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or lactose excipients in IP
21. Major surgery within 8 weeks prior to Week 0 Visit. Participants must have completely recovered from any previous surgery prior to Week 0 Visit
22. Prior heart or heart-lung transplants
23. Life expectancy of < 12 months (per PI determination)
24. Pregnant or breastfeeding females
25. At any time in the 30 days prior to the Screening Period received > 20 mg/day of prednisone (or equivalent) or started or changed the dose of a systemic corticosteroid. Participants receiving stable doses of ≤ 20 mg prednisone (or equivalent) in 30 days prior to the Screening Period are permitted in the study.
26. History of active malignancy within the past 5-years, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
27. History of clinically significant (as determined by the investigator) non-PAH related cardiac, endocrine, hematologic, hepatic, immune, metabolic, urologic, pulmonary, neurologic, neuromuscular, dermatologic, psychiatric, renal, and/or other disease that may limit participation in the study
28. Participation in another clinical trial involving intervention with another investigational drug or approved therapy for investigational use within 4 weeks prior to Week 0 Visit, or if the half-life of the previous product is known, within 5x the half-life prior to Week 0 Visit, whichever is longer
29. Participation in another clinical trial involving an investigational device within 4 weeks prior to Week 0 Visit
30. Unwillingness or inability to comply with the protocol- required procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline VO2 max | 24 weeks

SECONDARY OUTCOMES:
Change in VE/VCO2 slope (ventilatory efficiency) | 24 weeks
Change in cardiac output (CO) | 24 weeks
Change in cardiac index (CI) | 24 weeks
Change in stroke volume (SV) | 24 weeks
Change in mean pulmonary arterial pressure (mPAP) | 24 weeks
Change in pulmonary capillary wedge pressure (PCWP) | 24 weeks
Change in pulmonary vascular resistance (PVR) | 24 weeks
Change in pulmonary arterial compliance (PAC) | 24 weeks
Change in pulmonary arterial distensibility | 24 weeks
Change in CavO2 (arteriovenous O2 content difference) | 24 weeks
Change from baseline in RV SV, RV ESV, RV EDV, RV EF, RV SVI, RV ESVI and RV EDVI by cardiac magnetic resonance (MR) imaging | 24 weeks
Pharmacokinetic (PK) : Whole Blood Concentration of LAM-001 | 24 weeks
Change from baseline in 6MWD | 24 weeks
Change from baseline in WHO functional class | 24 weeks
Time to clinical worsening (from time of randomization until study discontinuation due to clinical worsening). | 24 weeks
Change from baseline in supplemental oxygen requirements | 24 weeks
Change from baseline in pulse oximetry | 24 weeks
Change from baseline in pulmonary function tests (PFTs) | 24 weeks
Exacerbations of underlying lung disease (WSPH Group-3) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No